CLINICAL TRIAL: NCT01126138
Title: A Randomized Phase III Study to Investigate the Efficacy and Safety of Docetaxel + Capecitabine vs. Vinorelbine + Capecitabine Followed by Capecitabine Alone as 1st Therapy on Locally Advanced and Metastatic Breast Cancer Patients.
Brief Title: Capecitabine (NX) Versus Docetaxel Plus Capecitabine (TX) as 1-line Chemotherapy on Metastatic Breast Cancer (MBC)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Prof. Binghe Xu, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML25241
Record Dates: First submitted 2010-05-18; First posted 2010-05-19 (Estimated); Last update posted 2011-05-04 (Estimated); Status verified 2010-05

CONDITIONS: Carcinoma, Invasive Ductal, Breast
Keywords: unresectable; locally advanced; metastatic; breast cancer
MeSH Terms: conditions — Carcinoma, Ductal, Breast; Neoplasm Metastasis; Breast Neoplasms | interventions — Vinorelbine; Capecitabine; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Other): Vinorelbine plus Capecitabine
  Interventions: Drug: Vinorelbine plus Capecitabine for 6 cycles, followed by Capecitabine
- Arm B (Other): Docetaxel plus Capecitabine
  Interventions: Drug: Docetaxel plus Capecitabine for 6 cycles, followed by Capecitabine

INTERVENTIONS:
Drug: Vinorelbine plus Capecitabine for 6 cycles, followed by Capecitabine — Capecitabine: 1,000 mg/m2 PO twice daily (day 1-14) Vinorelbine: 25 mg/m2 IV over 3 hours on day 1 and 8, every 3 weeks 21 days as one cycle and 6 cycles are required
  Arms: Arm A
Drug: Docetaxel plus Capecitabine for 6 cycles, followed by Capecitabine — Capecitabine: 1,000 mg/m2 PO twice daily (day 1-14), Docetaxel: 75 mg/m2 IV over 3 hours on day 1, every 3 weeks, 21 days as one cycle and 6 cycles are required.
  Followed by Capecitabine: 1,000 mg/m2 PO twice daily (day 1-14) 21 days as one cycle until progression or unacceptable toxicity
  Arms: Arm B

SUMMARY:
It is a phase III trial to explore the efficacy and safety of vinorelbine plus capecitabine (NX) and docetaxel plus capecitabine (TX) as first line treatment followed by capecitabine alone till Progressive Disease(PD). We plan to enroll 200 pts for limited budget and the non-inferior trend of the two curves is anticipated.

DETAILED DESCRIPTION:
We designed the randomized non-inferiority study. Main Inclusion& exclusion Criteria include: 1) Histologically or cytologically confirmed breast cancer with unresectable locally advanced and/or metastatic disease; 2) Untreated patients with unresectable locally advanced and/or metastatic disease; 3) with at least 1 lesion measurable by radiological method(RECIST criteria); 4) Karnofsky Performance Status(KPS)≥70; 5) normal Adequate hepatic, renal, and bone marrow function; 6) Life expectancy of at least 12 weeks; 7) No previous chemotherapy for metastatic breast cancer. Primary endpoint is Progression free survival(PFS), second endpoint are safety profiles (National Cancer Institute-Common Toxicity Criteria 3.0, NCI-CTC 3.0), overall survival and response rate. During Primary study treatment, Arm A: Capecitabine: 1,000 mg/m2 per ora(PO) twice daily (day 1-14), Vinorelbine 25 mg/m2 intravenous(IV) over 3 hours on day 1 and 8, every 3 weeks, 21 days as one cycle and 6-8 cycles are required; Arm B: Capecitabine: 1,000 mg/m2 PO twice daily (day 1-14), Docetaxel 75 mg/m2 IV over 3 hours on day 1, every 3 weeks, 21 days as one cycle and 6-8 cycles are required. Patients who are responding (complete or partial), or whose disease is stable followed by Capecitabine: 1,000 mg/m2 PO twice daily (day 1-14) 21 days as one cycle until progression or unacceptable toxicity

ELIGIBILITY:
Inclusion Criteria:

* Written and signed informed consent prior to beginning specific protocol procedures.
* Pathologically confirmed breast cancer and documented metastatic or locally advanced disease.

Measurable disease (RECIST criteria) - with at least 1 lesion measurable by radiological method

* KPS>=70
* Adjuvant and/or Neoadjuvant chemotherapy, including an anthracycline was permitted
* Hormone therapy for early-stage or metastatic breast cancer was permitted if hormonal receptor positive.
* Treatment with Herceptin for early-stage or metastatic breast cancer is permitted if HER2 positive
* Patients had to have concluded prior radiation therapy at least 14 days before enrollment.
* Laboratory requirements:

  * Hematology Absolute neutrophil count>=1,500 /μl; Platelets>=100,000 /μl; Hemoglobin>=10 g/dl
  * Liver function Total bilirubin<=2 times ULN ASAT (SGOT) and ALAT (SGPT)<=2.5 times UNL without liver metastasis or <=5.0 times if liver metastasis Glucose<=200 mg/dL
  * Renal function Serum creatinine<=140 mol/l
* Life expectancy of at least 12 weeks
* Patients must be accessible for treatment and follow-up.
* Patients should have recovered from the acute reversible effects of prior treatment. This generally means at least 3 weeks should have elapsed since prior chemotherapy, adjuvant or Neoadjuvant treatment. and at least 4 weeks since prior (radical) radiotherapy or major surgery

Exclusion Criteria:

* Women who are pregnant or breast feeding
* History of brain and/or leptomeningeal metastases
* Previous chemotherapy for metastatic breast cancer
* Past or current history of malignant neoplasm other than breast carcinoma, except for curatively treated non melanoma skin cancer, in situ carcinoma of the cervix or other cancer curatively treated and with no evidence of disease for at least 5 years
* Pre-existing neuropathy grade 1 according to the NCIC-CTC 3.0
* Psychiatric disorders or other conditions which would prevent pt. compliance
* Other serious illness or medical condition:

  * Congestive heart failure, or unstable angina pectoris, previous history of myocardial infarction within 6 month prior to study entry, uncontrolled hypertension as determined by the Investigator or high risk uncontrolled, arrhythmia.
  * History of significant neurological or psychiatric disorders including psychotic disorders, dementia of seizures that would prohibit the understanding and giving of informed consent.
  * Active uncontrolled infection.
  * Unstable peptic ulcer, unstable diabetes mellitus or other contraindication for the use of Corticosteroids.
* Inability to take and/or absorb oral medicine
* Prior treatment with an docetaxel and/or capecitabine and/or vinorbine
* Concurrent treatment with other experimental drugs, or participation in another clinical trial with any investigational drug within 30 days prior to study entry

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2010-07; Primary Completion 2015-05 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Progression free survival(PFS) | Up to 2 years until disease progression or death
  Progress free survival is defined as the time from first dose of test drug to the first recording of disease progression or the date of death in patients with no evidence of disease progression.
  In addition to hazard ratios and associated 95% confidence intervals, the results from these analyses will, for each treatment arm, also be summarized by Kaplan-Meier plots, medians and 95% confidence intervals.

SECONDARY OUTCOMES:
Safety Profiles | Up to 2 years until 28 days after last intake of study medication
  All adverse events occurring up to 28 days after last intake of study medication are to be recorded in the case report form. Safety profile will be analyzed by tabulating its occurring frequency and percentage per patient using NCI-CTC version 3.0. χ2 statistics will be used to test the differences in toxicities between the two treatment arms.
  SAEs will be reported according to ICH-GCP.
Overall Survival | Up to 3 years after last intake of study medication
  Survival will be measured from the date of first dose of test drug to the date of death (any cause) or to the date of last contact.
Response Rate | Up to 2 years until disease progression, unacceptable toxicity or death
  Tumor responses were assessed on the basis of Response Evaluation Criteria in Solid Tumours (RECIST) 1.1 at 6-week intervals then at 12-week intervals after disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: Binghe Xu, MD, Ph.D, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, China

REFERENCES:
- [Background] Sjostrom J, Blomqvist C, Mouridsen H, Pluzanska A, Ottosson-Lonn S, Bengtsson NO, Ostenstad B, Mjaaland I, Palm-Sjovall M, Wist E, Valvere V, Anderson H, Bergh J. Docetaxel compared with sequential methotrexate and 5-fluorouracil in patients with advanced breast cancer after anthracycline failure: a randomised phase III study with crossover on progression by the Scandinavian Breast Group. Eur J Cancer. 1999 Aug;35(8):1194-201. doi: 10.1016/s0959-8049(99)00122-7. PMID 10615229
- [Background] Ghosn M, Kattan J, Farhat F, Younes F, Gasmi J. Phase II trial of capecitabine and vinorelbine as first-line chemotherapy for metastatic breast cancer patients. Anticancer Res. 2006 May-Jun;26(3B):2451-6. PMID 16821631
- [Background] Welt A, von Minckwitz G, Oberhoff C, Borquez D, Schleucher R, Loibl S, Harstrick A, Kaufmann M, Seeber S, Vanhoefer U. Phase I/II study of capecitabine and vinorelbine in pretreated patients with metastatic breast cancer. Ann Oncol. 2005 Jan;16(1):64-9. doi: 10.1093/annonc/mdi024. PMID 15598940
- [Background] Chan A, Verrill M. Capecitabine and vinorelbine in metastatic breast cancer. Eur J Cancer. 2009 Sep;45(13):2253-65. doi: 10.1016/j.ejca.2009.04.031. Epub 2009 May 20. PMID 19464166
- [Result] O'Shaughnessy J, Miles D, Vukelja S, Moiseyenko V, Ayoub JP, Cervantes G, Fumoleau P, Jones S, Lui WY, Mauriac L, Twelves C, Van Hazel G, Verma S, Leonard R. Superior survival with capecitabine plus docetaxel combination therapy in anthracycline-pretreated patients with advanced breast cancer: phase III trial results. J Clin Oncol. 2002 Jun 15;20(12):2812-23. doi: 10.1200/JCO.2002.09.002. PMID 12065558